CLINICAL TRIAL: NCT02962050
Title: Delineating Physiologic Mechanisms of Swallowing Impairment and Decline in ALS
Brief Title: Delineating Swallowing Impairment and Decline in ALS
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201602098-N; R01NS100859 (NIH)
Record Dates: First submitted 2016-11-04; First posted 2016-11-11 (Estimated); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Respiratory Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ALS: Participants enrolled will complete the following tests: Videofluoroscopic Swallowing Study, Voluntary Peak Cough Flow Testing, lingual strength and endurance trials using the Iowa Oral Performance Instrument, reflexive cough testing, Pulmonary Function Testing; Eating Assessment Tool-10 (EAT-10), Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R), and the The Center for Neurologic Study Bulbar Function Scale (CNS-BFS).
  Interventions: Procedure: Videofluoroscopic Swallowing Study (VFSS); Device: Voluntary Peak Cough Flow Testing; Device: Iowa Oral Performance Instrument; Drug: Capsaicin Challenge; Device: Pulmonary Function Testing; Other: Eating Assessment Tool 10; Other: The Center for Neurologic Study Bulbar Function Scale

INTERVENTIONS:
Procedure: Videofluoroscopic Swallowing Study (VFSS) — Videofluoroscopic swallowing study will be performed to measure oropharyngeal swallowing
  Other Names: VFSS; X-Ray of Swallowing; Modified Barium Swallow Study
Device: Voluntary Peak Cough Flow Testing — Voluntary peak cough flow testing will be performed to determine the peak expiratory flow (PEF) and volume of air expelled (FEV1) during voluntary coughing.
Device: Iowa Oral Performance Instrument — The Iowa Oral Performance Instrument (IOPI) is a device that measures the peak pressure performance of lingual strength and endurance via the action of a bulb placed on the hard palate.
  Other Names: IOPI
Drug: Capsaicin Challenge — A capsaicin challenge with three randomized blocks of 0, 50, 100, 200, and 500 μM capsaicin. The capsaicin will be dissolved in a vehicle solution consisting of 80% physiological saline, and 20% ethanol. Participants will be given the instruction "cough if you need to" prior to capsaicin delivery.The solution will be administered automatically upon detection of an inspired breath and there will be a minimum of one minute between each trial. This is to test the reflexive cough testing for upper airway sensitivity and motor thresholds.
  Other Names: Reflexive Cough Testing
Device: Pulmonary Function Testing — Pulmonary Function testing will be performed using conventional methods and will include the following outcomes: forced vital capacity (FVC), maximum inspiratory pressure (MIP), and maximum expiratory pressure (MEP) expressed as a percentage of predicted values.
Other: Eating Assessment Tool 10 — The Eating Assessment Tool-10 will be used for participant reporting of swallowing system severity.
  Other Names: EAT 10
Other: The Center for Neurologic Study Bulbar Function Scale — The Center for Neurologic Studies Bulbar Function Scale (CNS-BFS) will be used to report bulbar function in study participants.
  Other Names: CNS-BFS

SUMMARY:
The purpose of this study is to 1) evaluate the discriminant ability of simple clinical markers to detect swallowing impairment in individuals with ALS, 2) develop and validate a minimally invasive clinical screening tool for use at multidisciplinary ALS clinics, and 3) determine the natural history of swallowing impairment and decline in ALS.

DETAILED DESCRIPTION:
This research study is being performed to determine screening tools or tests that are able to identify and track swallowing problems associated with Amyotrophic Lateral Sclerosis (ALS) over time. Also, this study will provide insight into the natural progression of swallowing impairment in persons with ALS over time.

Participants enrolled in this study will complete an evaluation at the University of Florida Aerodigestive Research Core laboratory located at Shands Hospital, Gainesville every three months. Each evaluation will take approximately 90 minutes. During these evaluations, a videofluoroscopy (X-ray of swallowing) examination, cough tests and questionnaires will be completed.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of probable or definite ALS

Exclusion Criteria:

* allergies to barium or capsaicin
* History of stroke
* Head and Neck Cancer
* Other disorder that might contribute to swallowing impairment
* Not enrolled in other research investigations that might impact swallowing
* Not pregnant

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with Amyotrophic Lateral Sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
Global Swallowing Function | Baseline, every 3 months through study completion, an average of 2 years.
  The DIGEST scale will be used by trained, blinded raters to assign ratings of safety to bolus trials. Both efficiency and safety will be assigned a score from 0-4 (more safe/efficient - less safe/efficient) and based on these ratings, will be given a total score ranging from 0-4 that captures their DIGEST rating.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Plowman, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - University of South Florida, Tampa, Florida